CLINICAL TRIAL: NCT03332823
Title: Community-based Mental Wellness Project for Adolescents and Adults: SME (Sharing, Mind, Enjoyment) Ambassadors Pilot Project
Brief Title: SME Ambassadors Pilot Project Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Council of Social Service (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, School of Nursing, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SPH-MHP-HKCSS02
Record Dates: First submitted 2017-10-29; First posted 2017-11-06 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Mental Well-being; Happiness
Keywords: Mental health; Mental well-being; Community-based engagement; Positive psychology; Public health approach
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SME Ambassadors training & program (Experimental): - SME Ambassadors will participate in train-the-ambassador workshops and provide voluntary services and promote mental well-being activities to vulnerable groups.
  Interventions: Behavioral: SME Ambassadors training & program

INTERVENTIONS:
Behavioral: SME Ambassadors training & program — * Two train-the-ambassador workshops: to train the ambassadors on positive thinking and understanding of adult mental health problem (in particular the mixed anxiety and depressive disorder) and mental well-being.
  * The trained SME ambassadors will provide voluntary services and promote mental well-being messages to vulnerable groups, such as ex-mental illness people, new arrivals, etc.

SUMMARY:
Aims: To enhance mental well-being of adults by creating a positive, happy and joyful environment in the community.

Targets: Adults aged 18-59 in Hong Kong.

Methods: SME Ambassadors Pilot Project will adopt the public health and family-focused approach, under the brand name of "Joyful@HK Campaign". Evidence-based and Evidence Generating approach with vigorous study design, both qualitative (e.g. focus groups) and quantitative (e.g. pre- and post- test), will be used to evaluate the overall programme effectiveness including follow-up of at least one month ("best science"). To ensure the practicability and sustainability of the community-based engagement project, we will engage community partners with strong track records of "best practice" to design, plan, and implement the intervention. This project will use innovative and integrated positive psychology and public health theories and methods to plan brief, simple, and cost-effective intervention.

Significance: By using "best science" in the design and evaluation of intervention programme, and the "best practice" of the partners' skills, experience and strong connection with service targets in the community, the intervention, if proven to be effective, for promoting sharing, mind and enjoyment and enhancing mental well-being can be further developed and widely disseminated to and adopted by the practitioners in the health and social service sectors for replication and improvement to benefit the whole population.

DETAILED DESCRIPTION:
SME Ambassadors Pilot Project is one of the six Community-based Mental Wellness Project for Adolescents and Adults, which aims at enhancing mental well-being of adolescents, adults and their families by creating a positive, happy and joyful environment in the community. The Project is funded by Health Care and Promotion Fund of Food and Health Bureau.

SME Ambassadors Pilot Project is organized by the Hong Kong Council of Social Service and led by School of Public Health, The University of Hong Kong(HKU). The project will organize two train-the-ambassador workshops to train 60-80 SME ambassadors on positive thinking and understanding of adult mental health problem (in particular the mixed anxiety and depressive disorder) and mental well-being.

The trained SME ambassadors will provide voluntary services and promote mental well-being messages to vulnerable groups, such as ex-mental illness people, new arrivals, etc.

The major subjects of the SME Ambassadors Pilot Project are 60-80 SME ambassadors who aged 18-59. 10-12 service providers from NGO service units (community partners) and 100-120 voluntary service recipients will also be involved in the study. Pre- and post-test evaluation will be used to evaluate the effectiveness of the intervention programme.

In the study, SME Ambassadors will be invited to complete questionnaires to measure their sharing, mind and enjoyment related behavioural indicators and invited to attend the focus group interviews to understand their experience during the programme; while community partners will be invited to attend individual interviews to collect their feedback and components on improving future community-based mental wellness programme.

Evaluation will be conducted during the programme implementation stage. The effectiveness of the intervention, as well as the level of participation and ratings for the intervention will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1) SME Ambassadors (major subjects):

* Adults who aged 18-59
* Chinese speaking
* Able to complete study questionnaires/ focus groups (2) Service recipients (which may include children/adolescents)
* Chinese speaking
* Able to complete study questionnaires/ focus groups (3) Community partners
* Service provider and participating NGO service units
* Chinese speaking
* Able to complete study questionnaires/ individual in-depth interviews

Exclusion Criteria:

* Those who cannot read Chinese
* Those who suffered from severe mental illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in participants' frequency of performing the suggested Sharing, Mind and Enjoyment (SME) related behaviours | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  The frequency of performing the SME (Sharing: share happy experience with others, help others, express care to others; Mind: recall the good memory, be grateful for what you already have, keep positive; Enjoyment: enjoy physical activity) related behaviours in the past 7 days will be assessed. The questions are rated 0-7 with 0 indicating none of this behavior happened in the past 7 days and 7 indicating this behavior happened every day in the past 7 days.

SECONDARY OUTCOMES:
Changes in personal happiness from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Personal happiness will be assessed by Subjective Happiness Scale (SHS). SHS was rated on 7-point scale with 1 indicating no happiness at all and 7 indicating extreme happiness. To score the scale, the 4th item will be coded reversely and mean of the 4 items will be computed.
Changes in mental well-being from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Mental well-being will be assessed by validated Chinese version of 7-item Warwick Edinburgh Well-being Scale. Each item ranges from 1 to 5 and the scale will be scored by first summing the score for each of the 7 items and then transforming the total score for each person according to a conversion table.
Changes in family relationship from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Self-perceived understanding, intimacy, and family communication will be assessed by three questions (rated 0-10).
Changes in individual and family health from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Self-perceived health, at the individual and family level will be assessed by two questions respectively (rated 0-10).
Changes in family happiness from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Self-perceived happiness, at the individual and family level will be assessed by two questions respectively (rated 0-10).
Changes in family harmony from baseline to three-month after baseline | T1: baseline; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Self-perceived family harmony will be assessed by a single question (rated 0-10).
Changes in knowledge and perception of mixed anxiety and depressive disorders | T1: baseline; T2: immediate post intervention; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Knowledge and perception of mixed anxiety and depressive disorders will be assessed by 4 questions (2 questions about understanding of symptoms, 1 about the intention of help seeking, 1 about support seeking from families) rated 0-10.
Satisfaction towards SME Ambassador Pilot Project | T2: immediate post intervention; T3: one-month follow-up after baseline; T4: three-month follow up after baseline
  Satisfaction towards programme will be assessed by conducting focus group and program evaluation measures (general satisfaction, self-perceived helpfulness and likely-to-recommend level) rated 0-10.
The social impact of the community-based engagement project | Up to four months
  The social impact of the community-based engagement project will be evaluated by conducting community stakeholders' in-depth interviews.
The process of community based intervention programme | Up to four months
  Assessed by a Process Evaluation on-site observation form, and a series of checklists including Resources input record sheet, Participants' attendance form, Programme rundown, Attendance record form, and NGOs' final report. The components of process evaluation, including context, reach, dose delivered, dose received, fidelity and recruitment will be assessed.
Outcomes of community engagement process | Up to four months
  Outcomes of community engagement process will be assessed by a self-designed questionnaire survey.

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, Principal Investigator — The University of Hong Kong
Locations (1):
- The Hong Kong Council of Social Service, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No